CLINICAL TRIAL: NCT03129763
Title: Perfusion Assessment With Indocyanine Green-SPY Angiography After Tissue Expander Filling for Optimization of Expansion Capsule Pressure
Brief Title: Perfusion Assessment With Indocyanine Green-SPY Angiography After Tissue Expander Filling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qing-FengLi Li,MD, MD, PhD, Professor, Head of Departement of Plastic and Reconstructive Surgery, Shanghai 9th People's Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2017]13
Record Dates: First submitted 2017-04-14; First posted 2017-04-26 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Tissue Expander Disorder
Keywords: SPY-ICG Angiography; Tissue Expander; Capsule Pressure; Blood Supply

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized controlled trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 60mmHg Group (Experimental): 60mmHg capsule pressure expansion. This pressure depends on the ideal capsule pressure that previous study given.
  Interventions: Behavioral: 60mmHg capsule pressure expansion
- 70mmHg Group (Experimental): 70mmHg capsule pressure expansion. This pressure gradient depends on the ideal capsule pressure that previous study given, and the regular expansion pressure in recent studies.
  Interventions: Behavioral: 70mmHg capsule pressure expansion
- 80mmHg Group (Experimental): 80mmHg capsule pressure expansion. This pressure gradient depends on the ideal capsule pressure that previous study given, and the regular expansion pressure in recent studies.
  Interventions: Behavioral: 80mmHg capsule pressure expansion
- 90mmHg Group (Experimental): 90mmHg capsule pressure expansion. This pressure gradient depends on the ideal capsule pressure that previous study given, and the regular expansion pressure in recent studies.
  Interventions: Behavioral: 90mmHg capsule pressure expansion
- 100mmHg Group (Experimental): 100mmHg capsule pressure expansion. This pressure gradient depends on the regular expansion pressure in recent studies.
  Interventions: Behavioral: 100mmHg capsule pressure expansion

INTERVENTIONS:
Behavioral: 60mmHg capsule pressure expansion — With a self-made apparatus composed of a spring-loaded sphygmomanometer and a disposable three-way pipe, the capsule pressure is measured. Increasing capsule pressure till 60mmHg.
  Arms: 60mmHg Group
Behavioral: 70mmHg capsule pressure expansion — With a self-made apparatus composed of a spring-loaded sphygmomanometer and a disposable three-way pipe, the capsule pressure is measured. Increasing capsule pressure till 70mmHg.
  Arms: 70mmHg Group
Behavioral: 80mmHg capsule pressure expansion — With a self-made apparatus composed of a spring-loaded sphygmomanometer and a disposable three-way pipe, the capsule pressure is measured. Increasing capsule pressure till 80mmHg.
  Arms: 80mmHg Group
Behavioral: 90mmHg capsule pressure expansion — With a self-made apparatus composed of a spring-loaded sphygmomanometer and a disposable three-way pipe, the capsule pressure is measured. Increasing capsule pressure till 90mmHg.
  Arms: 90mmHg Group
Behavioral: 100mmHg capsule pressure expansion — With a self-made apparatus composed of a spring-loaded sphygmomanometer and a disposable three-way pipe, the capsule pressure is measured. Increasing capsule pressure till 100mmHg.
  Arms: 100mmHg Group

SUMMARY:
The purpose of this study is to optimize the expansion pressure by compare different capsule pressures' effect, the blood supply of expanded skin is assessed by the Indocyanine Green-SPY Angiography.

DETAILED DESCRIPTION:
This is a randomized controlled trial that designed to optimize the tissue expander expanding method. All the patients were randomly divided into five groups, patients in different groups received an expansion weekly with different capsule pressure of 60mmHg, 70mmHg, 80mmHg, 90mmHg and 100mmHg respectively. Each patient received an expanding once a week, and a hemodynamic assessment of SPY-ICG angiography every two weeks. The total follow-up for each patient is 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 50 years;
* Expanding skin donor site at the face, neck, anterior chest wall or back;
* Implanted silicone expander of 100 to 600 ml in size; The quantitiy of normal saline in the tissue expander is more than the original volume, and less than double original volume.
* Need for further skin expansion; with previous regular expanding in hospital;

Exclusion Criteria:

* Iodine allergy; Indocyanine green allergy;
* Not fit for soft tissue expansion treatment;
* Evidence of infection, ischemia, ulcer or other pathological changes within the targeting area which defined as not suitable for expansion; or history of delayed healing, radiational therapy;
* Significant renal, cardiovascular, hepatic and psychiatric diseases;
* Significant medical diseases or infection (including but not limited to the carrier of hepatitis B virus or HIV)
* BMI >30;
* History of any hematological disease, including leukopenia , thrombocytopenia, or thrombocytosis;
* History of allogenic bone marrow transplantation;
* Long history of smoking;Evidence of malignant diseases or unwillingness to participate.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-07 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Expanded Skin Fluorescence Intensity Decrease Rate in Venous Phase (Unit per-second) | Baseline at visit 1, and post-expanding every two weeks in the follow-up.
  Engress Rate is one of the expanded skin perfusion relative quantitative index of Indocyanine Green-SPY Angiography. It is obtained by SPY-Q analysis, which represents the flow of expanded skin veins.

SECONDARY OUTCOMES:
Expanded Skin Fluorescence Intensity Increasion Rate in Arterial Phase (Unit per-second) | Baseline at visit 1, and post-expanding every two weeks in the follow-up.
  Ingress Rate is one of the expanded skin perfusion relative quantitative index of Indocyanine Green-SPY Angiography. It is obtained by SPY-Q analysis, which represents the flow of expanded skin arteries.
Expanded Skin Fluorescence Intensity Increasion in Arterial Phase (Unit) | Baseline at visit 1, and post-expanding every two weeks in the follow-up.
  Ingress is one of the expanded skin perfusion relative quantitative index of Indocyanine Green-SPY Angiography. It is obtained by SPY-Q analysis, which represents the absolute value of expanded skin fluorescence intensity increasion in arterial phase.
Expanded Skin Fluorescence Intensity Decrease in Venous Phase (Unit) | Baseline at visit 1, and post-expanding every two weeks in the follow-up.
  Engress is one of the expanded skin perfusion relative quantitative index of Indocyanine Green-SPY Angiography. It is obtained by SPY-Q analysis, which represents the absolute value of expanded skin fluorescence intensity decrease in venous phase.

CONTACTS AND LOCATIONS:
Overall Officials: Qingfeng Li, MD; PhD, Study Director — Shanghai Ninth People's Hospital, Affliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Ninth People's Hospital, Affliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China